CLINICAL TRIAL: NCT03189472
Title: Remotely-supervised Transcranial Direct Current Stimulation (tDCS) for At-home Treatment of Fatigue and Cognitive Slowing in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-00486
Record Dates: First submitted 2017-06-05; First posted 2017-06-16 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active tDCS (Experimental)
  Interventions: Device: Active tDCS
- sham tDCS (Sham Comparator)
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — low amplitude direct currents to induce changes in cortical excitability. tDCS produces current intensities in the brain orders of magnitude below other stimulation techniques such as transcranial magnetic stimulation (TMS) or electroconvulsive therapy (ECT)
  Other Names: Remotely Supervised Transcranial Direct Current Stimulation
  Arms: active tDCS
Device: Sham tDCS — The device will be programmed to deliver either active or sham tDCS (all study personnel and participants will be blinded), and operated with unlock codes provided by the study technician daily to release one session
  Arms: sham tDCS

SUMMARY:
This is a double-blind randomized controlled pilot study to test the effects of Remotely-Supervised (RS)-tDCS using a dorsolateral prefrontal cortex montage to ameliorate fatigue and cognitive slowing in PD.

Fatigue and slowed thinking are very prevalent symptoms in people with Parkinson's disease (PD). To date there are no concrete effective treatment available for either symptom. This study will test transcranial direct current stimulation (tDCS) to ameliorate fatigue and slowed thinking in PD. tDCS is a noninvasive brain stimulation technique that is low-cost, relatively safe, and reproducible when conducted in repeat clinic visits.

Following procedures for our validated protocol, participants will receive training on the use of study tDCS device and pre configured laptop computer. The device will be programmed to deliver either active or sham tDCS (all study personnel and participants will be blinded), and operated with unlock codes provided by the study technician daily to release one session. Once trained, and following an initial in-clinic baseline tDCS tolerability test and initial treatment session, participants will use the equipment to complete the remaining sessions from their home using our tele medicine platform. Remote supervision will be provided using HIPAA secure online video conference with the study technician following clearly-defined operational procedures. Participants will be monitored to determine if any predefined "stop" criteria are met using VSee software, a telemedicine software. Additionally, Team Viewer software will allow study technicians to troubleshoot any computer issues, to initiate the video conference on behalf of participants, and to remotely supervise the entire tDCS session.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD confirmed by neurologist;
* Parkinson fatigue scale binary coding scoring a score of > 7;
* Able to understand the informed consent process and provide consent to participate in the study
* Has stable and continuous access to internet service at home compatible with the study laptop (Wi-Fi or ethernet cable)
* Adequate internet capacity for remote monitoring, as tested by http://www.speedtest.net/)
* Subjects who are stable in their PD medication for 2 or more weeks prior to enrollment.

Exclusion Criteria:

* Visual, auditory and motor deficits that would prevent full ability to understand study instructions or operate the tDCS device or study laptop, as judged by treating neurologist or study staff
* Current chronic headaches or migraines. In addition, if a subject has had a change in the rate or severity of head pressure, headache, or migraine in the past two weeks, they are excluded.
* History of significant head trauma (e.g., brain injury, brain surgery) or medical device implanted in the head (such as Deep Brain Stimulator) or in the neck (such as a Vagus Nerve Stimulator)
* Any skin disorder/sensitive skin (e.g., eczema, severe rashes, blisters, open wounds, burn including sunburns, cuts or irritation, or other skin defects) which compromise the integrity of the skin at or near stimulation locations where electrodes are placed
* Serious uncontrolled medical condition (e.g., cancer or acute myocardial infarction)
* Alcohol or other substance use disorder
* Hoehn and Yahr score >3
* Pregnant or breastfeeding
* History of dementia or Montreal Cognitive Assessment (MoCA) score <20
* Not capable of passing the neuropsychology /computer and tDCS aptitude test
* Unable to tolerate discomfort from the tDCS tolerability stimulation test

Ages: 35 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Number of participants having completed 80% sessions | 5 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Drummond, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States